CLINICAL TRIAL: NCT04132999
Title: Positive Airway Pressure for the Treatment of the Obstructive Sleep Apnea Syndrome in Children With Down Syndrome (Stage 2)
Brief Title: PAP for Children With DS and OSAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Children's Hospital Medical Center, Cincinnati (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20230780; R61HL151253-01 (NIH); R33HL151253 (NIH)
Record Dates: First submitted 2019-10-10; First posted 2019-10-21 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Down Syndrome; Obstructive Sleep Apnea
Keywords: Down Syndrome; Obstructive Sleep Apnea; PAP; Positive Airway Pressure
MeSH Terms: conditions — Down Syndrome; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: family-informed intervention (INT) vs standard clinical care (CON).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family-informed intervention (INT) (Active Comparator): Multiple face-to-face visits, telephone calls and-person visits with the PAP psychologist and team.
  Interventions: Behavioral: Family-informed intervention
- Standard Clinical Care (Active Comparator): Support which is given as part of the standard clinical care for patients who are currently prescribed PAP.
  Interventions: Behavioral: Standard Clinical Care

INTERVENTIONS:
Behavioral: Family-informed intervention — Multiple face-to-face visits, telephone calls and-person visits with the PAP psychologist and team
  Arms: Family-informed intervention (INT)
Behavioral: Standard Clinical Care — Support which is given as part of the standard clinical care for patients who are currently prescribed PAP.
  Arms: Standard Clinical Care

SUMMARY:
Determine the efficacy of family-informed intervention (INT) vs standard clinical care over a period of twelve months in children with obstructive sleep apnea and Down Syndrome.

DETAILED DESCRIPTION:
Evaluate the effect of PAP adherence on quality of life, neurobehavioral, and healthcare utilization in children with DS and OSAS. It is being hypothesized that, irrespective of study arm, increased PAP adherence will be associated with better quality of life, neurobehavioral, and healthcare utilization outcomes.

Evaluate the effect of PAP adherence in children with DS and OSAS on patient-centered outcomes and family-relevant outcomes identified during the R61 phase of this research. It is being hypothesized that irrespective of study arm, increased PAP adherence will be associated with better patient-centered outcomes, and family-relevant outcomes identified during the first year of this research.

Determine the efficacy of INT vs. CON in promoting PAP adherence. It is being hypothesized that that children receiving INT will show significantly increased objectively-measured PAP adherence at 6 months compared with those receiving CON (Aim 4A). As a secondary aim (4B), it will be evaluated whether the improved adherence is maintained over 12 months. It is being hypothesized that participants initially randomized to the INT arm will have better adherence at 12 months compared to those in the CON arm.

Use mixed methods during the randomized controlled trial to identify family perceptions, such as empowerment and self-efficacy, regarding PAP use in youth with OSAS and DS. It is being hypothesized that INT-PAP will be associated with more positive perceptions compared to CON.

ELIGIBILITY:
Inclusion Criteria:

* Clinical referral for PAP initiation to treat OSAS
* Ages 6-18 years
* Children are able to cooperate with testing
* Naive to PAP treatment

Exclusion Criteria:

* Major illnesses, such as leukemia or severe cyanotic congenital heart disease listed for cardiac transplant.
* Family planning to move out of the city within the next year
* Children in foster care
* Child with previously treated with PAP
* Caregivers who do not speak English well enough to complete behavioral and performance measures.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 86 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Effect of PAP adherence on quality of life and neurobehavioral outcomes | Baseline, 6 months, and 12 months
  PedsQL score and measures of executive functioning will be compared in the 2 groups. PedsQL is a 5-point scale ranging from 0-4 (0 = Never, 4 = Always).
Efficacy of INT-PAP in promoting PAP adherence | 6 months, and 12 months
  Adherence to PAP expressed as percentage of nights used, and minutes of usage on nights used.
Efficacy of CON in promoting PAP adherence | 6 months, and 12 months
  Adherence to PAP expressed as percentage of nights used, and minutes of usage on nights used.
Effect of PAP adherence in children with DS and OSAS on patient-centered outcomes and family-relevant outcomes identified during the R61 phase of this research | Baseline, 6 months, and 12 months
  Patient-centered outcomes and family-relevant outcomes - identified during the R61 phase of the study (Stage 1) - will be compared between the intervention and control groups. These are qualitative measures, and require interviews and further analysis to be established.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Miami, Miami, Florida
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xanthopoulos MS, Byars K, Meinzen-Derr J, Ebensen A, Xiao R, Heubi C, Gurbani NS, Ishman SL, Bradford R, Hicks S, Redline S, Tapia IE. Standard medical care versus enhanced interdisciplinary care for implementation of positive airway pressure in youth with Down syndrome: a randomised controlled trial protocol. BMJ Open. 2025 Nov 23;15(11):e110990. doi: 10.1136/bmjopen-2025-110990. PMID 41285506